CLINICAL TRIAL: NCT03231007
Title: Saving Babies' Lives Project Impact and Results Evaluation: a Mixed Methodology Study
Acronym: SPiRE
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Collaborators: Somerset NHS Foundation Trust (Other); Royal Devon and Exeter NHS Foundation Trust (Other); University Hospital Plymouth NHS Trust (Other); Royal United Hospital Bath NHS Trust (Other); North Bristol NHS Trust (Other); Liverpool Women's NHS Foundation Trust (Other); St Helens & Knowsley Teaching Hospitals NHS Trust (Other); Countess of Chester NHS Foundation Trust (Other); University Hospitals of Morecambe Bay NHS Trust (Other); Barnsley Hospital NHS Foundation Trust (Other); Doncaster And Bassetlaw Hospitals NHS Foundation Trust (Other); York Teaching Hospitals NHS Foundation Trust (Other); Hull University Teaching Hospitals NHS Trust (Other Government); Mid Yorkshire Teaching NHS Trust (Other); Oxford University Hospitals NHS Trust (Other); Gateshead Health NHS Foundation Trust (Other); North Cumbria University Hospitals NHS Trust (Other); Sherwood Forest Hospitals NHS Foundation Trust (Other); Manchester University NHS Foundation Trust (Other Government); Birmingham Women's NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Dr Alexander Heazell, Professor of Obstetrics, University of Manchester
Other Study IDs: R04666
Record Dates: First submitted 2017-07-06; First posted 2017-07-27 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Stillbirth
MeSH Terms: conditions — Stillbirth | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Innovators: Maternity units that implemented the Care Bundle to the highest level (according to an NHS survey in 2015) are categorised as 'Innovators'.
  Interventions: Other: Questionnaire
- Early Adopters: Maternity units that implemented the Care Bundle to the second-highest level (according to an NHS survey in 2015) are categorised as 'Early Adopters'.
  Interventions: Other: Questionnaire
- Late Adopters: Maternity units that implemented the Care Bundle to the third-highest level (according to an NHS survey in 2015) are categorised as 'Late Adopters'.
  Interventions: Other: Questionnaire
- Low Adopters: Maternity units that implemented the Care Bundle to the fourth-highest level (according to an NHS survey in 2015) are categorised as 'Low Adopters'.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A structured questionnaire will be administered to maternity service users. Another structured questionnaire will be administered to maternity healthcare professionals, and another to Organisational Leads (e.g. Clinical Directors at each site).

SUMMARY:
The study is a multicentre evaluation of maternity care delivered through the Saving Babies' Lives care bundle using both quantitative and qualitative methodologies. The study will be conducted in twenty NHS Hospital Trusts from six NHS Strategic Clinical Networks totalling approximately 100,000 births. It involves participation by both service users and care providers.

To determine the impact of the care bundle on pregnancy outcomes, birth data and other clinical measures will be extracted from maternity databases and case-note audit from before and after implementation. Additionally, this study will employ questionnaires with organisational leads and review clinical guidelines to assess how resources, leadership and governance may affect implementation in diverse hospital settings. The cost of implementing the care bundle, and the cost per stillbirth avoided, will also be estimated as part of a health economic analysis. The views and experiences of service users and service providers towards maternity care in relation to the care bundle will be also be sought using questionnaires.

This study will provide practice-based evidence to advance knowledge about the processes that underpin successful implementation of the care bundle so that it can be further developed and refined. This has the potential to translate into substantial improvements in the rate of late stillbirth in the UK should the care bundle be proved effective.

DETAILED DESCRIPTION:
Reducing stillbirth and early neonatal death is a national priority. Best practice and key evidence indicates this is potentially achievable through application of four key interventions within routine maternity care delivered as NHS England's Saving Babies' Lives care bundle. However, adoption of the care bundle by UK maternity services is still in its infancy and there is significant variation in the degree of implementation between and within units. The effectiveness of the care bundle, when implemented as a package, in reducing stillbirth and service delivery has not yet been evaluated. This study aims to evaluate the impact of implementing the care bundle on UK maternity services and perinatal outcomes.

ELIGIBILITY:
Inclusion Criteria for Maternity Service Users:

* Women who received their antenatal care, delivered and were discharged from the same maternity unit
* Women who have given birth after 28 weeks of gestation

Exclusion Criteria for Maternity Service Users:

* Maternal age ≤ 16 years
* Individuals who cannot understand/not fluent in English (to enable consent without interpreter)
* Multiple pregnancy
* Fetuses known to have any congenital or severe structural abnormalities
* Home births

Inclusion Criteria for Maternity Healthcare Professionals:

* Midwives working before and after implementation of the care bundle (including antenatal ward, antenatal clinic, community-based staff, antenatal assessment unit and labour ward)
* Community midwives working before and after implementation of the care bundle
* Sonographers working before and after implementation of the care bundle
* Junior doctors working before and after implementation of the care bundle
* Consultant obstetricians working before and after implementation of the care bundle
* Clinical Directors and Heads of Midwifery working before and after implementation of the care bundle

Exclusion Criteria for Maternity Healthcare Professionals:

- Staff who were employed after the care bundle was implemented

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Postnatal service users who have received antenatal care and given birth in one of the 20 study sites.
  Healthcare professionals who are involved in delivering maternity care in one of the 20 study sites.
Sampling Method: Non-Probability Sample
Enrollment: 4952 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Stillbirths | 1st April 2012-1st October 2017
  All stillbirths (singletons and multiples). Stillbirths will be defined according to the UK definition as the death of a baby before or during birth after 24 weeks of gestation.

SECONDARY OUTCOMES:
Term, normally formed singleton stillbirths (antepartum and intrapartum). | 1st April 2012-1st October 2017
  This excludes issues of preterm birth and major mortality and morbidity associated with congenital anomalies.
Preterm births | 1st April 2012-1st October 2017
Babies' gestation | 1st April 2012-1st October 2017
Number of reported incidents | 1st April 2012-1st October 2017
Admission to NICU | 1st April 2012-1st October 2017
Antenatal triage numbers | 1st April 2012-1st October 2017
Emergency caesarean deliveries | 1st April 2012-1st October 2017
Induced deliveries | 1st April 2012-1st October 2017
Birthweight | 1st April 2012-1st October 2017
Birthweight centile | 1st April 2012-1st October 2017
  Using GROW-Centile software
Spontaneous deliveries | 1st April 2012-1st October 2017
Caesarean deliveries | 1st April 2012-1st October 2017
Instrumental deliveries | 1st April 2012-1st October 2017

OTHER OUTCOMES:
Process Outcome - Care Bundle Element 1 (Smoking in Pregnancy): Proportion of women smoking at delivery | 10th July 2017-31st August 2017
Process Outcome - Care Bundle Element 1 (Smoking in Pregnancy): Proportion of women offered carbon monoxide (CO) test | 10th July 2017-31st August 2017
Process Outcome - Care Bundle Element 1 (Smoking in Pregnancy): Proportion of women accepting CO test | 10th July 2017-31st August 2017
Process Outcome - Care Bundle Element 1 (Smoking in Pregnancy): Proportion of women referred to smoking cessation | 10th July 2017-31st August 2017
Process Outcome - Care Bundle Element 1 (Smoking in Pregnancy): Proportion of women ceasing smoking between booking and delivery | 10th July 2017-31st August 2017
Process Outcome - Care Bundle Element 1 (Smoking in Pregnancy): Proportion of women referred to smoking cessation with a positive CO test | 10th July 2017-31st August 2017
Process Outcome - Care Bundle Element 2 (Small for Gestational Age Detection): Proportion of SGA singletons detected prior to delivery | 1st April 2012-1st October 2017
Process Outcome - Care Bundle Element 2 (Small for Gestational Age Detection): Proportion of all singletons with growth charts in notes | 1st April 2012-1st October 2017
Process Outcome - Care Bundle Element 2 (Small for Gestational Age Detection): Proportion of SGA pregnancies with estimated fetal weight (EFW) plotted on growth chart | 1st April 2012-1st October 2017
Process Outcome - Care Bundle Element 2 (Small for Gestational Age Detection): Proportion of SGA pregnancies with symphysis fundal height (SFH) plotted on growth chart | 1st April 2012-1st October 2017
Process Outcome - Care Bundle Element 2 (Small for Gestational Age Detection): Proportion of SGA pregnancies with EFW correctly plotted on growth chart | 1st April 2012-1st October 2017
Process Outcome - Care Bundle Element 2 (Small for Gestational Age Detection): Proportion of babies identified as SGA during pregnancy that were appropriate for gestation age (AGA) at birth (false positives) | 1st April 2012-1st October 2017
Process Outcome - Care Bundle Element 2 (Small for Gestational Age Detection): Proportion of babies identified as AGA during pregnancy that were SGA at birth (false negatives) | 1st April 2012-1st October 2017
Process Outcome - Care Bundle Element 2 (Small for Gestational Age Detection): Proportion of pregnancies with customised growth chart | 1st April 2012-1st October 2017
Process Outcome - Care Bundle Element 2 (Small for Gestational Age Detection): Birthweight centile at last scan (by EFW measurement) | 1st April 2012-1st October 2017
Process Outcome - Care Bundle Element 2 (Small for Gestational Age Detection): Number of third trimester growth scans | 1st April 2012-1st October 2017
Process Outcome - Care Bundle Element 3 (Patient Information Provision and Reduced Fetal Movements Management): Proportion of women receiving RFM leaflet | 1st April 2012 until 1st October 2017
Process Outcome - Care Bundle Element 3 (Patient Information Provision and Reduced Fetal Movements Management): Proportion of women with RFM managed | 1st April 2012 until 1st October 2017
Process Outcome - Care Bundle Element 3 (Patient Information Provision and Reduced Fetal Movements Management): Number of triage women presenting with RFM on at least one occasion | 1st April 2012 until 1st October 2017
Process Outcome - Care Bundle Element 3 (Patient Information Provision and Reduced Fetal Movements Management): Proportion of women with RFM who had scan | 1st April 2012 until 1st October 2017
Process Outcome - Care Bundle Element 3 (Patient Information Provision and Reduced Fetal Movements Management): Proportion of women with RFM who had FH monitoring | 1st April 2012 until 1st October 2017
Process Outcome - Care Bundle Element 3 (Patient Information Provision and Reduced Fetal Movements Management): Gestation of baby at RFM episodes | 1st April 2012 until 1st October 2017
Process Outcome - Care Bundle Element 3 (Patient Information Provision and Reduced Fetal Movements Management): Number of growth scans due to RFM | 1st April 2012 until 1st October 2017
Process Outcome - Care Bundle Element 3 (Patient Information Provision and Reduced Fetal Movements Management): Time to scan from reporting RFM | 1st April 2012 until 1st October 2017
Process Outcome - Care Bundle Element 3 (Patient Information Provision and Reduced Fetal Movements Management): Number of RFM episodes per pregnancy according to checklist | 1st April 2012 until 1st October 2017
Process Outcome - Care Bundle Element 4 (Effective Fetal Monitoring During Labour): Proportion of deliveries where both buddy and stickers used | 1st April 2012 until 1st October 2017
Process Outcome - Care Bundle Element 4 (Effective Fetal Monitoring During Labour): Proportion of staff completing annual CTG training | 1st April 2012 until 1st October 2017
Process Outcome - Care Bundle Element 4 (Effective Fetal Monitoring During Labour): Proportion of pregnancies where escalation protocol was used | 1st April 2012 until 1st October 2017
Process Outcome - Care Bundle Element 4 (Effective Fetal Monitoring During Labour): Number of babies therapeutically cooled | 1st April 2012 until 1st October 2017
Economic Outcome - Equipment required | 10th July 2017-31st August 2017
  (e.g. CO test kits)
Economic Outcome - Staff time required | 10th July 2017-31st August 2017
  (e.g. to conduct additional scans)
Economic Outcome - Antenatal triage numbers | 10th July 2017-31st August 2017
Economic Outcome - Number of triage women presenting with RFM on at least one occasion | 10th July 2017-31st August 2017
Economic Outcome - Emergency caesarean deliveries | 10th July 2017-31st August 2017
Economic Outcome - Induced deliveries | 10th July 2017-31st August 2017
Economic Outcome - Caesarean deliveries | 10th July 2017-31st August 2017
Economic Outcome - Number of third trimester growth scans | 10th July 2017-31st August 2017
Economic Outcome - Number of growth scans due to RFM | 10th July 2017-31st August 2017
Economic Outcome - Number of antenatal CTGs due to RFM | 10th July 2017-31st August 2017
Economic Outcome - Length of stay in NICU | 10th July 2017-31st August 2017
Economic Outcome - Length of stay in hospital | 10th July 2017-31st August 2017

CONTACTS AND LOCATIONS:
Locations (20):
- United Kingdom (20):
  - Barnsley Hospital NHS Foundation Trust, Barnsley
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - North Bristol NHS Trust, Bristol
  - North Cumbria University Hospitals NHS Trust, Carlisle
  - Countess of Chester Hospital NHS Foundation Trust, Chester
  - Doncaster and Bassetlaw Hospitals NHS Foundation Trust, Doncaster
  - Royal Devon & Exeter NHS Foundation Trust, Exeter
  - Gateshead Health NHS Foundation Trust, Gateshead
  - Oxford University Hospitals NHS Trust, Headington
  - Hull and East Yorkshire Hospital NHS Trust, Hull
  - University Hospitals of Morecambe Bay NHS Foundation Trust, Kendal
  - Liverpool Women's NHS Foundation Trust, Liverpool
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - Plymouth Hospital NHS Trust, Plymouth
  - St Helens and Knowsley Teaching Hospitals NHS Trust, Prescot
  - Sherwood Forest Hospitals NHS Foundation Trust, Sutton in Ashfield
  - Taunton and Somerset NHS Foundation Trust, Taunton
  - The Mid Yorkshire Hospitals NHS Trust, Wakefield
  - York Teaching Hospital NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Office of National Statistics. Characteristics of birth 1, England and Wales, 2013. London: ONS, 2014.
- [Background] Flenady V, Wojcieszek AM, Middleton P, Ellwood D, Erwich JJ, Coory M, Khong TY, Silver RM, Smith GCS, Boyle FM, Lawn JE, Blencowe H, Leisher SH, Gross MM, Horey D, Farrales L, Bloomfield F, McCowan L, Brown SJ, Joseph KS, Zeitlin J, Reinebrant HE, Cacciatore J, Ravaldi C, Vannacci A, Cassidy J, Cassidy P, Farquhar C, Wallace E, Siassakos D, Heazell AEP, Storey C, Sadler L, Petersen S, Froen JF, Goldenberg RL; Lancet Ending Preventable Stillbirths study group; Lancet Stillbirths In High-Income Countries Investigator Group. Stillbirths: recall to action in high-income countries. Lancet. 2016 Feb 13;387(10019):691-702. doi: 10.1016/S0140-6736(15)01020-X. Epub 2016 Jan 19. PMID 26794070
- [Background] Manktelow BN, S.L., Seaton SE, Hyman-Taylor P, Kurinczuk JJ, Field DJ. MBRRACE-UK Perinatal Mortality Surveillance Report, UK Perinatal Deaths for Births from Janurary to December 2014. Leicester: The Infant Mortality and Morbidity Studies, Department of Health Sciences, University of Leicester, 2016.
- [Background] Draper ES, K.J., Kenyon S (Eds) on behalf of MBRRACE-UK, MBRRACE-UK Perinatal Confidential Enquiry. Term, singleton, normally formed, antepartum stillbirth. Leicester: The Infant Mortality and Morbidity Studies, Department of Health Sciences, Univesity of Leicester. 2015.
- [Background] Widdows K, Roberts SA, Camacho EM, Heazell AEP. Stillbirth rates, service outcomes and costs of implementing NHS England's Saving Babies' Lives care bundle in maternity units in England: A cohort study. PLoS One. 2021 Apr 19;16(4):e0250150. doi: 10.1371/journal.pone.0250150. eCollection 2021. PMID 33872334
- [Background] Gardosi J, Madurasinghe V, Williams M, Malik A, Francis A. Maternal and fetal risk factors for stillbirth: population based study. BMJ. 2013 Jan 24;346:f108. doi: 10.1136/bmj.f108. PMID 23349424
- [Background] Marufu TC, Ahankari A, Coleman T, Lewis S. Maternal smoking and the risk of still birth: systematic review and meta-analysis. BMC Public Health. 2015 Mar 13;15:239. doi: 10.1186/s12889-015-1552-5. PMID 25885887
- [Background] RCOG Green-Top Guideline 31: The Investigation and Management of the Small-for-Gestational Ages Fetus. Royal College of Obstetricians and Gynaecologists, 2013.
- [Background] Alfirevic Z, Devane D, Gyte GM. Continuous cardiotocography (CTG) as a form of electronic fetal monitoring (EFM) for fetal assessment during labour. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD006066. doi: 10.1002/14651858.CD006066. PMID 16856111
- [Derived] Widdows K, Reid HE, Roberts SA, Camacho EM, Heazell AEP. Saving babies' lives project impact and results evaluation (SPiRE): a mixed methodology study. BMC Pregnancy Childbirth. 2018 Jan 30;18(1):43. doi: 10.1186/s12884-018-1672-x. PMID 29378526

DOCUMENTS (1):
  • Study Protocol (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT03231007/Prot_000.pdf